CLINICAL TRIAL: NCT04966481
Title: Palbociclib and Cetuximab Versus Cetuximab Monotherapy for Patients With CDKN2A-altered, HPV-unrelated Head and Neck Squamous Cell Carcinoma Who Experienced Disease Progression on a PD-1/L1 Inhibitor: A Multicenter, Open-Label, Randomized Phase 3 Trial
Brief Title: Palbociclib and Cetuximab Versus Cetuximab Monotherapy for Patients With CDKN2A-altered, HPV-unrelated Head and Neck Squamous Cell Carcinoma Who Experienced Disease Progression on a PD-1/L1 Inhibitor
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry); The Joseph Sanchez Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202108203
Record Dates: First submitted 2021-07-07; First posted 2021-07-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: HPV-unrelated Head and Neck Squamous Cell Carcinoma
MeSH Terms: interventions — palbociclib; Cetuximab

STUDY DESIGN:
Intervention Model Description: These patients will be randomized on a 2:1 basis to Arm 1 (palbociclib + cetuximab, n=54) or Arm 2 (cetuximab alone, n=27). Patients will be stratified at randomization to balance the proportion of patients in each arm with:
  1. previous exposure to a platinum agent (cisplatin or carboplatin given to treat recurrent or metastatic disease, or as a component of multimodality therapy for newly diagnosed locally advanced, non-metastatic HNSCC),
  2. previous exposure to cetuximab (given as a component of multimodality therapy for newly diagnosed locally advanced, non-metastatic HNSCC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Palbociclib + Cetuximab (Experimental): * Palbociclib by mouth 125 mg/daily on Days 1-21 of each 28 day cycle
  * Cetuximab: Initial dose 400mg/m^2 intravenous (IV); Subsequent doses 250 mg/m^2 IV, weekly
  Interventions: Drug: Palbociclib; Drug: Cetuximab
- Arm 2: Cetuximab (Active Comparator): -Cetuximab: Initial dose 400mg/m^2 intravenous (IV); Subsequent doses 250 mg/m^2 IV, weekly
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Palbociclib — Administered on an outpatient basis
  Other Names: Ibrance
  Arms: Arm 1: Palbociclib + Cetuximab
Drug: Cetuximab — Given intravenously over approximately 60 minutes
  Other Names: Erbitux

SUMMARY:
This multicenter, open-label, randomized phase 3 trial will determine if palbociclib and cetuximab (Arm 1) improves overall survival (OS) in comparison to cetuximab monotherapy (Arm 2) in patients with CDKN2A-altered, HPV-unrelated recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) who experienced disease progression on a PD-1/L1 inhibitor (given as monotherapy or in combination with other therapy).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed RM-HNSCC that is HPV-unrelated disease; defined as SCC of the oral cavity, larynx, or hypopharynx and p16 negative SCC of the oropharynx or p16 negative non-cutaneous SCC unknown primary of the neck.
* CDKN2A loss-of-function (LOF) alteration: mutation or homozygous deletion described on genomic sequencing report.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam, per RECIST 1.1.
* Disease progression on a PD-1/L1 inhibitor-containing regimen (given as monotherapy or in combination with other therapy).
* Received no more than three lines of prior therapy for RM-HNSCC.
* At least 18 years of age.
* ECOG performance status ≤ 1.
* Normal bone marrow and organ function as defined below:

  * Hemoglobin ≥ 8 g/L
  * Absolute neutrophil count ≥ 1,000/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 3 x institutional upper limit of normal (IULN)
  * AST(SGOT)/ALT(SGPT) ≤ 5 x IULN (for cases involving liver metastases, AST/ALT ≤ 10 x IULN)
  * Serum creatinine < 3 x IULN or creatinine clearance > 30 mL/min by Cockcroft-Gault
* The effects of palbociclib and cetuximab on the developing human fetus are unknown. For this reason and because CDK 4/6 inhibitors are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 3 months days after completion of the study
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior treatment with cetuximab for recurrent or metastatic disease (however, prior cetuximab given as a component of multimodality therapy for newly diagnosed, locally advanced, non-metastatic HNSCC is allowable).
* Prior treatment with a CDK4/6 inhibitor for RM-HNSCC.
* Rb (retinoblastoma) loss: mutation or homozygous deletion described on genomic sequencing report.
* Currently receiving any other investigational agents.
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 1 year before registration and the patient has no evidence of recurrent/persistent disease.
* Patients with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT scan) during the screening period
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib or other agents used in the study (excluding cetuximab).
* Prior grade 3 or 4 (per CTCAE 5.0) hypersensitivity reaction to cetuximab.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* QTc >500 msec (using Bazette formula).
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended. Recommend exclusion of specific ART agents based on predicted drug-drug interactions (i.e. for sensitive CYP3A4 substrates, concurrent strong CYP3A4 inhibitors (ritonavir and cobicistat) or inducers (efavirenz) should be contraindicated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Through completion of follow-up (estimated to be 15 months)
  -Defined as the time from the date of treatment to the date of death, censored at the last follow-up otherwise.

SECONDARY OUTCOMES:
Overall response rate (ORR) - (complete response + partial response) | Through completion of treatment (estimated to be 12 weeks)
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Duration of response (DoR) | Through completion of treatment (estimated to be 12 weeks)
  -The duration of response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 15 months)
  * Defined as the days from the date of treatment start to progression or death. The alive patients without progression are censored at the last follow-up.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. ): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Frequency of adverse events | From start of treatment through 30 days after completion of treatment (estimated to be 16 weeks)
  -Will be measured by CTCAE v. 5.0
Dose delivery as measured by percent of full doses given over time | Through completion of treatment (estimated to be 12 weeks)
Correlate CCND1 and PIK3CA alterations with efficacy endpoints | Through completion of follow-up (estimated to be 15 months)
  Tailored Next Generation Sequencing Report (performed before trial enrollment) will be collected to tabulate additional somatic genomic alterations to be used to correlate with efficacy endpoints.
Changes in genomic alterations of tumor | At baseline and at time of progression (estimated to be 15 months)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Saint Luke's Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Medical Center, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu